CLINICAL TRIAL: NCT06600113
Title: Evaluating Effectiveness of Different Educational Methods on the Anxiety of Children Undergoing Anaesthesia - a Randomized Controlled Trial
Brief Title: Effect of Educational Intervention on Children's Anxiety
Acronym: MINA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iceland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: UI-2022-MINA
Record Dates: First submitted 2024-02-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Health Literacy; Anesthesia; Anxiety; Fear; Attitude; Child Behavior; Health Knowledge, Attitudes, Practice
Keywords: Children; Game; Anesthesia; Health literacy
MeSH Terms: conditions — Anxiety Disorders; Behavior; Child Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Game playing (Experimental): Children play a specially designed educational game within one week of their medical procedure. The game informs the child what to expect at the day of the procedure and teaching coping strategies
  Interventions: Other: Education and teaching of coping strategies
- Story telling (Active Comparator): Children are read an illustrated story by their parent within one week of their medical procedure. The story informs the child what to expect at the day of the procedure and teaching coping strategies
  Interventions: Other: Education and teaching of coping strategies
- Usual care (No Intervention): These children get the usual care, information from their parents or doctor before the medical procedure

INTERVENTIONS:
Other: Education and teaching of coping strategies — the intervention consists of patient education for children, the same content delivered through either an educational game and storytelling
  Arms: Game playing; Story telling

SUMMARY:
The aim of this randomized controlled trial is to evaluate the effectiveness of an educational health game intervention for children undergoing anesthesia from the perspective of children's anxiety. Participants are divided into three groups: one plays an educational game, another gets similar educational material (story) on a website and the third receives usual care. Anxiety will be evaluated with a standard assessment tool at the medical centre and parents answer questionnaires about themselves and their child. The study is an important step into innovation in the field of patient education where computer games are used to disseminate information, teach salvation and promote faith in the child's own ability and courage. The study will provide important information on children's anxiety for anaesthesia and what the effects of the computer game are compared to other educational methods.

DETAILED DESCRIPTION:
This study is a randomized controlled trial. This study will evaluate the effectiveness of an educational health game intervention for children undergoing anesthesia from the perspective of children's anxiety. The data will be collected from children (4-8 years old) and their parent or guardian at four different time points: the baseline, post1, post-2 and post 3-intervention.

The sample size was calculated by statistician using power calculations. According to the calculations, the targeted sample size is in total 150 children (50 per each arm) in Finland and Iceland.

Participants are recruited from daycare surgery wards in university hospitals or hospitals where children undergo various procedures under anesthesia. The recruitment will be agreed separately with the hospital and hospital workers.

Data will be collected in four different time points.

1. Before the intervention, baseline. Questionnaires for parent: the child's temperament is measured with Child Behaviour Questionnaire (CBQ) (Rothbart et al 2001), the anxiety of parent is measured with the State-trait Anxiety Inventory (STAI, trait part) (Spielberger, 1983) and background information of the child and parents.
2. After the baseline questionnaires children are randomized to three groups. Group A: plays an educational mobile game, Group B: similar educational material on a website than in the health game, and Group C: the usual care (receives information from the health personnel) for preparation for the anesthesia.
3. At the hospital. Questionnaire for parent: Parents answers the anxiety of parent (STAI, state part). Nurse observes child's anxiety in hospital using The Modified Yale Preoperative Anxiety Scale, mYPAS short form, (mYPAS-SF) (Jenkins et al. 2014) in the waiting room before the anesthesia (post 1) while the child is prepared for anesthesia and right before the induction of anesthesia (post 2). Nurse 2 also observes weather the child is particularly crying or calm when waking up. The nurse will collect information from the child's medical records for the study, such as the procedure the child has had and the reason for the procedure, premedication etc.
4. After the anesthesia (post 3) Questionnaire for parent: 2-4 days after the operation questions regarding the experience of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing anesthesia for medical procedure

Exclusion Criteria:

* Does not understand Icelandic/Finnish

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative anxiety of children | Through study completion, twice a day of surgery: In the waiting room before anesthesia and just before induction of anesthesia.
  Anxiety is measured with short version of the modified Yale Preoperative Anxiety Scale (mYPAS-SF) with observational scores from 22.9, minimal anxiety, to 100, maximal anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Brynja Ingadottir, Ph.D, Principal Investigator — University of Iceland
Locations (1):
- Laeknastofur Akureyrar, Akureyri, Iceland

IPD SHARING:
Plan to Share IPD: No